CLINICAL TRIAL: NCT07040449
Title: Stress Trajectories and Anhedonia in Adolescence Research Study
Acronym: STAARS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 24-1236; R01MH136102 (NIH)
Record Dates: First submitted 2025-06-18; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Anhedonia; Stress Response; Adolescent Development
MeSH Terms: conditions — Anhedonia; Fractures, Stress | interventions — Psychological Tests

STUDY DESIGN:
Intervention Model Description: 1. The Trier Social Stress Test for Children (TSST-C)-- Psychosocial stress procedure in which the individual tells a story for 5 minutes in front of two neutral judges and performs mental arithmetic in front of the judges for 5 minutes.
  2. The Montreal Imaging Stress Task (MIST) -- Psychosocial stress procedure consisting of completing sections of mental arithmetic that are 5.5 minutes in length, during which the individual receives neutral and negative evaluative feedback about their performance relative to their peers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adolescent Teenagers (Experimental): Participants aged 13-15 (approximately Tanner pubertal stage 2-4) at study entry.
  Interventions: Behavioral: Montreal Imaging Stress Task; Behavioral: Trier Social Stress Test for Children

INTERVENTIONS:
Behavioral: Montreal Imaging Stress Task — Psychosocial stress procedure consisting of completing sections of mental arithmetic that are 5.5 minutes in length, during which the individual receives neutral and negative evaluative feedback about their performance relative to their peers.
Behavioral: Trier Social Stress Test for Children — Psychosocial stress procedure in which the individual tells a story for 5 minutes in front of two neutral judges and performs mental arithmetic in front of the judges for 5 minutes.

SUMMARY:
This project will examine how multiple biological measures from the brain and the body's stress response system contribute to anhedonia (the loss of pleasure) in adolescence. The goal of this project is to see if it is possible to combine these biological measures to describe different patterns of activity in the brain and body that adolescents may have in response to stress.

The main question this study aims to answer is whether different patterns of activity in the brain and body are related to whether adolescents develop anhedonia and how high or low levels of anhedonia are over time.

This study will enroll 192 adolescents who are between 13 and 15 years. Adolescents will complete tasks three times: at the beginning of the study, 10 months after that, and then 10 months after that. In total, they will be part of the study for 20 months. At each time, adolescents will complete surveys, provide samples of spit to measure hormones and provide pictures of their brain to measure brain activity, participate in mildly stressful tasks, and complete different activities that measure how they think. The investigators will also ask each adolescent's parent or legal guardian to answer some surveys about themselves and their child.

DETAILED DESCRIPTION:
Participants will complete tasks at 3 timepoints (Baseline, 10-Months, and 20-Months). Some tasks will be in-person, while others will be virtual.

The assessments being administered at all three timepoints are:

* Psychological measures (self-report, completed remotely): Anticipatory and Consummatory Interpersonal Pleasure Scale (ACIPS), Mood and Feelings Questionnaire short version (MFQ), Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Distress and Anxiety, PROMIS Psychological Stress Experiences, Snaith-Hamilton Pleasure Scale (SHAPS), Temporal Experience of Pleasure Scale (TEPS)
* Cognitive (researcher administered, conducted in-person): NIH Cognitive Toolbox
* Brain Imaging via functional magnetic resonance imaging (fMRI)
* Physiological (researcher administered, conducted in-person): Heart Rate Variability (HRV), Photoplethysmography (PPG), Impedance Cardiography (ICG), Pre-Ejection Period (PEP), Salivary Cortisol

Additionally, the following will be administered at each respective timepoint:

Baseline Assessment (Month 0):

Self-Report, Remote Questionnaires: demographic survey, address history survey, Protocol for Responding to & Assessing Patients' Assets, Risks & Experiences (PRAPARE), Pediatric Adverse Childhood Experiences and Related Life-events Screener (PEARLS) Cognitive (researcher administered, conducted in-person: Wechsler Abbreviated Scale of Intelligence Second Version (WASI-II) Psychological interview: Kiddie Schedule for Affective Disorders and Schizophrenia (KSADS)

Time 2 (10-Months) Juvenile Victimization Questionnaire (JVQ) (self-report, completed remotely)

Time 3 (20-Months) Psychological interview: Abbreviated Kiddie Schedule for Affective Disorders and Schizophrenia (KSADS)

ELIGIBILITY:
Inclusion Criteria:

* Age 13-15 years old at study entry
* Ability to understand and sign an assent form
* Meets study hearing and vision requirements

Exclusion Criteria:

* Current use of antipsychotic medication
* Current use of medications that would interfere with cardiovascular or endocrine assessments
* Metal in the body or other MRI exclusion
* Central nervous system disorder or brain injury that could confound brain imaging evaluations
* Presence of a medical condition that would interfere with cardiovascular or endocrine assessments
* Impaired intellectual functioning
* Diagnosed with a neurodevelopmental disability

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 192 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2030-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Anhedonia as assessed by the SHAPS | Baseline, 10-months, 20-months
  The Snaith-Hamilton Pleasure Scale (SHAPS) is a 14-item measure used to assess anhedonia. Each item has four answer responses: "strongly agree" (1 point), "agree" (2 points), "disagree" (3 points), and "strongly disagree" (4 points). The sum of these responses is taken to find the total score, which ranges from 0-56 with higher scores indicating more overall anhedonia.
Percent signal change during the MIST | Baseline, 10-Months, 20-Months
  During the MIST, research participants complete mental arithmetic with the intermittent reception of neutral and negative evaluative feedback. The percent signal change of the fronto-limbic region of the brain will be analyzed during the MIST task. Higher percent signal change in these regions would indicate higher levels of activation when stressed. Percent signal change ranges between 1% to 5%.
Endocrine (cortisol) response during the TSST | Baseline, 10-Months, 20-Months
  The Trier Social Stress Test for Children (TSST-C) -- a social stressor involving story telling in front of two neutral judges, preparation time and a cognitive stressor involving mental arithmetic is used to elicit physiological stress responses. The combination of stressors offers high levels of social-evaluative threat. Cortisol is collected through a saliva sample of passive drool a total of 5 times throughout the visit at 15-minute intervals. The higher the cortisol is found to be, the higher the stress response to the task.
Endocrine (cortisol) response during the MIST | Baseline, 10-Months, 20-Months
  During the MIST, research participants complete mental arithmetic with the intermittent reception of neutral and negative evaluative feedback. Cortisol is collected through a saliva sample collected via cotton swab a total of 6 times throughout the visit at 15-minute intervals. The higher the cortisol is found to be, the higher the stress response to the task.
Sympathetic and Parasympathetic nervous system ECG activation or heart rate variability (HRV) during a psychosocial stressful task (Trier Social Stress Test - TSST) | Baseline, 10-Months, 20-Months
  The Trier Social Stress Test for Children (TSST-C) -- a social stressor involving story telling in front of two neutral judges, preparation time and a cognitive stressor involving mental arithmetic is used to elicit physiological stress responses. The combination of stressors offers high levels of social-evaluative threat. Throughout the task, heart rate is measured to determine baseline resting state and HRV. HRV is the difference in the milliseconds between each heartbeat. The higher the HRV, the more the nervous system is activated during the task. The level of HRV indicates the participant's nervous system response to stress.

SECONDARY OUTCOMES:
Anhedonia as assessed by the ACIPS | Baseline, 10-months, 20-months
  The Anticipatory and Consummatory Interpersonal Pleasure Scale (ACIPS) assesses the ability to experience social pleasure. It contains 17-items scored on a 6-point Likert scale ranging from "very false for me" (1) to "very true for me" (6). The sum of these responses is taken to find the total score, which ranges from 17-102 with higher scores indicating lower capacity to experience or anticipate social pleasure.
Anhedonia as assessed by the TEPS | Baseline, 10-months, 20-months
  The Temporal Experience of Pleasure Scale (TEPS) is an 18-item measure used to assess anhedonia. It is scored on a 6-point Likert scale ranging from "very false for me" (1) to "very true for me" (6). The sum of these responses is taken to find the total score, which ranges from 18-108 with higher scores indicating more overall anhedonia.

CONTACTS AND LOCATIONS:
Overall Officials: Aysenil Belger, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Danielle Roubinov, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with National Institute of Mental Health (NIMH) policy, all individual-level data will be shared through the NIMH National Data Archive (NDA).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available to the public after the conclusion of the study and the publication of the manuscripts.
Access Criteria: Access to the data is limited to individuals who meet the following data access eligibility criteria as described on the NIMH NDA website:
  1. Research Need
  2. Electronic Research Administration (eRA) Commons Account
  3. Institutional Association
  4. Active Federal-Wide Assurance (FWA)
  5. NDA Account
URL: https://nda.nih.gov/